CLINICAL TRIAL: NCT05682495
Title: A Bioequivalence Study of HR20031 Tablet in Healthy Subjects
Brief Title: A HR20031 BE Study on Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HR20031-101
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: There will be two independent cohorts of subjects who will each receive two treatments (high dose strength and low dose strength), and each treatment will be followed by 72 hours of blood sampling for pharmacokinetic assessments, with safety and tolerability. In each cohort approximately 42 healthy subjects will be randomized to receive treatment with IP to complete at least 36 evaluable subjects.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ARM A：SHR3824 10 mg+ SP2086 100 mg+ Metformin 500 mg XR*2 (Experimental)
  Interventions: Drug: ARM A
- ARM B：HR20031 FDC 10/100/1000 mg (Experimental)
  Interventions: Drug: ARM B
- ARM C：SHR3824 10 mg+ SP2086 100 mg+ Metformin 500 mg XR*2 (Experimental)
  Interventions: Drug: ARM C
- ARM D：SHR3824 5 mg*2+ SP2086 50 mg*2+ Metformin 500 mg XR*3 (Experimental)
  Interventions: Drug: ARM D
- ARM E：HR20031 FDC 5/50/750 mg*2 (Experimental)
  Interventions: Drug: ARM E
- ARM F：SHR3824 5 mg*2+ SP2086 50 mg*2+ Metformin 500 mg XR*3 (Experimental)
  Interventions: Drug: ARM F

INTERVENTIONS:
Drug: ARM A — Subjects will receive treatment SHR3824 10 mg+ SP2086 100 mg+ Metformin 500 mg XR*2 followed by 7 days washout ，then receive treatment SHR3824 10 mg+ SP2086 100 mg+ Metformin 500 mg XR*2 followed by 7 days washout and then receive treatment HR20031 FDC 10/100/1000 mg.
  Arms: ARM A：SHR3824 10 mg+ SP2086 100 mg+ Metformin 500 mg XR*2
Drug: ARM B — Subjects will receive treatment HR20031 FDC 10/100/1000 mg followed by 7 days washout ，then receive treatment SHR3824 10 mg+ SP2086 100 mg+ Metformin 500 mg XR*2 followed by 7 days washout and then receive treatment SHR3824 10 mg+ SP2086 100 mg+ Metformin 500 mg XR*2.
  Arms: ARM B：HR20031 FDC 10/100/1000 mg
Drug: ARM C — Subjects will receive treatment SHR3824 10 mg+ SP2086 100 mg+ Metformin 500 mg XR*2 followed by 7 days washout ，then receive treatment HR20031 FDC 10/100/1000 mg followed by 7 days washout and then receive treatment SHR3824 10 mg+ SP2086 100 mg+ Metformin 500 mg XR*2.
  Arms: ARM C：SHR3824 10 mg+ SP2086 100 mg+ Metformin 500 mg XR*2
Drug: ARM D — Subjects will receive treatment SHR3824 5 mg*2+ SP2086 50 mg*2+ Metformin 500 mg XR*3 followed by 7 days washout ，then receive treatment SHR3824 5 mg*2+ SP2086 50 mg*2+ Metformin 500 mg XR*3 followed by 7 days washout and then receive treatment HR20031 FDC 5/50/750 mg*2.
  Arms: ARM D：SHR3824 5 mg*2+ SP2086 50 mg*2+ Metformin 500 mg XR*3
Drug: ARM E — Subjects will receive treatment HR20031 FDC 5/50/750 mg*2 followed by 7 days washout ，then receive treatment SHR3824 5 mg*2+ SP2086 50 mg*2+ Metformin 500 mg XR*3 followed by 7 days washout and then receive treatment SHR3824 5 mg*2+ SP2086 50 mg*2+ Metformin 500 mg XR*3.
  Arms: ARM E：HR20031 FDC 5/50/750 mg*2
Drug: ARM F — Subjects will receive treatment SHR3824 5 mg*2+ SP2086 50 mg*2+ Metformin 500 mg XR*3 followed by 7 days washout ，then receive treatment HR20031 FDC 5/50/750 mg*2 followed by 7 days washout and then receive treatment SHR3824 5 mg*2+ SP2086 50 mg*2+ Metformin 500 mg XR*3.
  Arms: ARM F：SHR3824 5 mg*2+ SP2086 50 mg*2+ Metformin 500 mg XR*3

SUMMARY:
The purpose of this study is to assess the bioequivalence between HR20031 FDC tablet and co-administration of SHR3824 tablets, SP2086 tablets and metformin XR tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial, and fully understand the content, process and possible adverse reactions of the trial. Must be able to communicate with the investigator, understand and comply with all study requirements;
2. Male or female subjects aged 18 to 45 (including 18 and 45);
3. Weigh at least 50 kg (for male) and 45 kg (for female), respectively, and have a body mass index (BMI) ≥ 19 and ≤28 kg/m2. BMI = weight (kg)/[height (m)]2;
4. Fasting plasma glucose in the range of 3.9-6.1 mmol/L.

Exclusion Criteria:

1. Subject (include their fere) have pregnancy plan from 2 weeks prior to dose administration to follow-up period and refuse to use effective form of birth control;
2. Those who have a positive urine drug screen or have a history of drug abuse;
3. Excessive smoking (≥ 5 cigarettes/day);
4. History of alcoholism or regular alcohol consumption within 1 month before screening, that is, drinking more than 14 units of alcohol per week (1 unit = 360 mL of beer with 5% alcohol or 45 mL of spirits with 40% alcohol or 150 mL of wine with 12% alcohol)
5. Subjects who took any beverage or food containing grapefruit, xanthine, caffeine, or alcohol within 48 hours before dosing or other factors which affect drug absorption, distribution, metabolism, excretion, etc
6. Subjects with medical conditions that may affect the absorption, distribution, metabolism, and excretion of the drug or impair adherence to the drug as judged by the investigator or deemed inappropriate by the investigator;
7. Viral hepatitis (including hepatitis B and C), AIDS antibody, and Treponema pallidum antibody screening are positive;
8. Clinical laboratory tests have clinically significant abnormalities;
9. Abnormal ECG has clinical significance;
10. Other clinical findings before screening show clinical significance for the following diseases (including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, Mental or cardiovascular disease);
11. History of allergy to test drugs, allergic constitution (multiple drug and food allergies);
12. Subjects who undergone any surgery within 3 months before screening, have not recovered from surgery, or have plans to surgery or hospitalization during the trial;
13. Donate blood or lose a lot of blood (>400mL) within three months before screening;
14. Subjects with a history of severe hypoglycaemia;
15. Subjects with a history of recurrent urinary tract infection or/and genital fungal infection;
16. Participated in the drug clinical trial and have taken drug or within three months before taking the research drug;
17. Take any prescription drugs, any vitamin products or herbal medicines within 14 days before screening or take any over-the-counter drugs within 1 month before screening;
18. Exposure to metformin and/or SGLT2 inhibitors such as dapagliflozin, empagliflozin, canagliflozin, ertugliflozin, and DPP-IV inhibitors such as sitagliptin, saxagliptin, linagliptin, or vildagliptin within 1 month before screening.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics parameters of SHR3824 in the fed state: Cmax | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of SP2086 in the fed state: Cmax | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of Metformin in the fed state: Cmax | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of SHR3824 in the fed state: AUC0-t | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of SP2086 in the fed state: AUC0-t | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of Metformin in the fed state: AUC0-t | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of SHR3824 in the fed state: AUC0-inf (if applicable) | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of SP2086 in the fed state: AUC0-inf (if applicable) | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of Metformin in the fed state: AUC0-inf (if applicable) | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15

SECONDARY OUTCOMES:
Pharmacokinetics parameters of SP2086A in the fed state: Cmax | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of SP2086A in the fed state: AUC0-t | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of SP2086A in the fed state: AUC0-inf (if applicable) | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of SHR3824 in the fed state: Tmax | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of SP2086 and SP2086A in the fed state: Tmax | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of Metformin in the fed state: Tmax | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of SHR3824 in the fed state: CL/F | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of SP2086 and SP2086A in the fed state: CL/F | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of Metformin in the fed state: CL/F | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of SHR3824 in the fed state: t1/2 | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of SP2086 and SP2086A in the fed state: t1/2 | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
Pharmacokinetics parameters of Metformin in the fed state: t1/2 | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15
The incidence and severity of adverse events/serious adverse events | Based on pre-dose, 0.25-72 hours post-dose sampling times on Day 1 and Day 8 and Day 15

CONTACTS AND LOCATIONS:
Locations (1):
- Jinan Central Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided